CLINICAL TRIAL: NCT00399100
Title: Is it Possible to Treat Cyanide Poisoning With HBO?
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: 01-277/99
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2006-11

CONDITIONS: Carbon Monoxide Poisoning From Fire Accidents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: HBO - hyperbaric oxygen treatment

SUMMARY:
People who has been in a fire accident have been shown often to be cyanide poisoned as well as poisoned with carbon monoxide(CO). According to recommendations from the Danish Health Agency people who are CO poisoned must be treated with hyperbaric oxygen (HBO). We want to see if HBO treatment can also treat cyanide poisoning.

The hypothesis is that as cyanide binds the same place in the mitochondria as CO cyanide will be detached from the mitochondria like CO and diffuse back to the blood.This way it will be easier to treat with hydroxycobalamin.

ELIGIBILITY:
Inclusion Criteria:

* Going to receive HBO treatment for carbon monoxide poisoning from fire accidents

Exclusion Criteria:

* Under 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-11 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Lawson-Smith, Doctor, Principal Investigator — Rigshospitalet HOC, Trykkammeret
Locations (1):
- Lab. for hyperbar medicin, afs. 4092, Anæstesi og Operationsklinikken, HOC, Rigshospitalet, København Ø, Denmark